CLINICAL TRIAL: NCT06136936
Title: A Multicenter, Exploratory, Randomized, Double-Arm, 4-week Study to Evaluate the Overall Effects of Treatment With Abbreviated CT-156 in People With Schizophrenia
Brief Title: A Study to Evaluate the Overall Effects of Treatment With Abbreviated CT-156 in People With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Click Therapeutics, Inc. (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Device Feasibility
Other Study IDs: CT-156-C-001
Record Dates: First submitted 2023-11-03; First posted 2023-11-18 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Software as a Medical Device (SaMD); Smartphone app
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- CT-156 (Active Comparator): Study app investigational treatment for adult patients diagnosed with schizophrenia.
  Interventions: Device: CT-156-C-001
- CT-156 + UXR (Experimental): Study app investigational treatment for adult patients diagnosed with schizophrenia with up to five in-patient visits with three interviews for UXR (user experience research) arm.
  Interventions: Device: CT-156-C-001

INTERVENTIONS:
Device: CT-156-C-001 — CT-156 is a digital therapeutic (DTx) under development to treat patients 18 years of age and older with a diagnosis of schizophrenia under standard of care therapy who are on antipsychotic medication and not currently experiencing acute hallucinations or delusions.

SUMMARY:
An exploratory, double-arm, 4-week study to explore the feasibility and acceptability of abbreviated treatment with CT-156 for people with Schizophrenia.

DETAILED DESCRIPTION:
The purpose of the proposed study is to evaluate the overall effects of use of an abbreviated version of CT-156 (the Study App) in participants aged 18 years or older with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* A participant will be eligible for entry into the study if all of the following criteria are met:

  1. Willing and able to provide written informed consent to participate in the study, attend study visits, and comply with study-related requirements and assessments.
  2. Is an adult at least 18 years of age at the time of informed consent.
  3. Fluent in written and spoken English, confirmed by ability to read and understand the informed consent form.
  4. Lives in the United States.
  5. Meets diagnostic criteria for a primary diagnosis of schizophrenia as defined in the International Classification of Diseases, Eleventh Edition (ICD-11) or Diagnostic Statistical Manual, Fifth Edition (DSM-5) for at least 6 months prior to screening.
  6. Has outpatient treatment status at the time of screening, with no psychiatric inpatient hospitalization within 13 weeks (3 months) prior to screening.
  7. Is currently prescribed at least one typical and/or atypical antipsychotic medication, and has been on the same antipsychotic medication(s) for at least 13 weeks (3 months) prior to randomization (Day 1). Dose adjustments are permitted during the study as outlined in the respective package insert(s).
  8. Has an average score of >2 in at least 2 domains of Understanding and communicating, Getting Along with People, Life Activities - Household, or Participation in Society on the World Health Organization Disability Assessment Schedule 2.0 (WHO-DAS 2.0).
  9. Participant is the only user of an iPhone with iPhone operating system (iOS) version 14 or later or a smartphone with an Android operating system (OS) version 11 or later and agrees to download and use the digital mobile application as required by the protocol.
  10. Is willing and able to receive SMS text messages and push messages on their smartphone.
  11. Is the owner of and has regular access to an email address.
  12. Has regular access to the internet via cellular data plan and/or wi-fi.
  13. Has stable housing and has remained at the same residence for at least 13 weeks (3 months) prior to screening, and does not anticipate housing changes for the duration of the study.
  14. Understands the use of the Study App during the screening period and at the Baseline Visit, per investigator judgment.

Exclusion Criteria:

* A participant will not be eligible for study entry if any of the following criteria are met:

  1. Has acute prominent positive symptoms that, in the opinion of the investigator, would preclude effective engagement with the app
  2. Is currently receiving or has received concomitant therapy, defined as individual or group-based structured treatment (e.g., Cognitive Behavioral Therapy, Social Skills Training, Motivational Interviewing, or Vocational/Occupational Therapy), within 6 months (26 weeks) prior to screening per investigator assessment.
  3. Is currently treated with more than two antipsychotic medications (including more than 2 dosage forms).
  4. Is currently treated with clozapine, or was treated with clozapine within 5 years of the Screening Visit.
  5. Meets ICD-11 or DSM-5 criteria for diagnoses not under investigation that will impact compliance to the protocol, including schizophreniform, schizoaffective, or psychosis non-specific disorders (post-traumatic stress disorder [PTSD], bipolar disorder, major depressive disorder, developmental disorders).
  6. Meets ICD-11 or DSM-5 criteria for a current episode of depression, mania or hypomania.
  7. Meets ICD-11 or DSM-5 criteria for a current substance or alcohol use disorder (excluding caffeine and nicotine) within 26 weeks (6 months) of the Screening Visit. Diagnoses classified as in sustained remission are permitted.
  8. In the investigator's opinion, currently needs or will likely require prohibited concomitant medications and/or therapy during the study.
  9. Is at risk for suicide, as defined by any of the following:

     1. A "yes" response to either item 4 or 5 on the C-SSRS Suicidal Ideation Items within the last 13 weeks (3 months) prior to screening or at the Baseline Visit.
     2. A "yes" response on the C-SSRS Suicidal Behavior Items within the last 26 weeks (6 months) prior to screening or at the Baseline Visit.
     3. In the opinion of the investigator, presents a serious risk of suicide.
  10. Has participated in another clinical study (interventional or observational) in the last 26 weeks (6 months).
  11. Has previously participated in study CT-155-C-001, CT-155-C-002, CT-155-C-003, CT-155-P-00x, or CT-155-A-001.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2024-01-18 (Actual); Study Completion 2024-02-22 (Actual)

PRIMARY OUTCOMES:
Number of days used | Day 0 to Week 4
  Number of days the Study App is opened out of total days of treatment
Number of times Study App is opened | Day 0 to Week 4
  Number of times the Study App is opened during the treatment period
Number of tasks completed | Day 0 to Week 4
  Number of assigned tasks completed during the treatment period
Length of time in App | Day 0 to Week 4
  Length of each App-use session

CONTACTS AND LOCATIONS:
Overall Officials: Shaheen Lakhan, Study Director — Click Therapeutics
Locations (1):
- Click Therapeutics, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No